CLINICAL TRIAL: NCT05617833
Title: Safety of Combined Therapy With Erythropoietin and Melatonin for Very Preterm Infants With Intraventricular Hemorrhage (SCEMPI)
Brief Title: Safety of Erythropoietin and Melatonin for Very Preterm Infants With Intraventricular Hemorrhage
Acronym: SCEMPI
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00301237; R01HD104673-01A1 (NIH)
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Intraventricular Hemorrhage of Prematurity
Keywords: SCEMPI; Erythropoietin; Melatonin; preterm infants; Intraventricular Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MLT+EPO (Experimental): Melatonin 3 mg/mL oral syringe enterally every evening. Dose will be divided in half and administered at evening cares.
  High dose epoetin alfa epbx recombinant (1000 units/kg) syringe subcutaneously or intravenously every 48 hours for 10 doses.
  Low dose epoetin alfa-epbx recombinant (400 units/kg) subcutaneously or intravenously three times weekly on Monday, Wednesday, and Friday until age 33-6/7wk.
  Interventions: Combination Product: MLT+EPO
- Placebo (Placebo Comparator): Placebo oral syringe enterally every evening.
  Placebo syringe IV every 48 hours for 10 doses.
  Placebo subcutaneously or intravenously three times weekly on Monday, Wednesday, and Friday until age 33-6/7wk.
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: MLT+EPO — Melatonin component will be a daily dose of 30 mg/kg enteral administered in the evening in a split dose given at cares/feedings. EPO component is a two-stage regimen with high dose EPO (1000 U/kg/dose q 48 hrs ± 2hr subcutaneously or intravenously) for 10 doses followed by maintenance dose EPO (400 U/kg/dose q Monday, Wednesday, Friday subcutaneously or intravenously) to 33-6/7wk. Maintenance EPO dosing will begin on the day closest to completing the high dose series.
  Arms: MLT+EPO
Other: Placebo — Placebo enteral and IV
  Arms: Placebo

SUMMARY:
Very preterm infants are prone to numerous medical complications with lifelong impact. Amongst the most serious are significant intraventricular hemorrhage (sIVH) and the subsequent progression to posthemorrhagic hydrocephalus (PHH). Currently, the only treatment for PHH is surgery, most commonly with shunts that are prone to malfunction across the lifespan. Preclinical data show that melatonin (MLT) and erythropoietin (EPO), when administered in a sustained dosing regimen, can prevent the hallmarks of progression from early postnatal sIVH to subsequent PHH. The investigators will perform a Phase I, single institution, randomized, double-blind trial for very preterm infants with sIVH to define a safe combination dose of MLT and EPO. A maximum of 60 very preterm neonates with sIVH will be enrolled, treated through 33w6/7d, and followed to 37w6/7d. Neonates will be randomized 3:1 between MLT+EPO and placebo, with all receiving standard of care. The primary endpoint is a composite serious adverse event (SAE)/dose limiting toxicity (DLT). The investigators hypothesize that the MLT+EPO SAE/DLT rate will not be higher than the placebo rate. Secondary outcomes will be rate of co-morbidities of preterm birth. Exploratory data, collected to guide design of future clinical trials for efficacy, will include serial neuro-imaging metrics acquired from clinical images, serial neonatal neurodevelopmental examinations, serum and urine MLT and EPO levels, and liquid biomarkers. Successful implementation of this initial safety trial will provide essential data to guide the next stage of clinical trials to test if sustained MLT+EPO treatment can reduce the need for surgical intervention, and avoid the lifelong burden of shunted hydrocephalus.

ELIGIBILITY:
Inclusion Criteria:

1. Neonatal intensive care unit (NICU) inpatients born at >22 and <32 weeks gestation (born after 22w-6/7 and before or on 31-6/7 week GA)
2. sIVH within the first 21 days from birth, defined as at least unilateral grade II on head ultrasound (HUS) performed within 18 days of enrollment
3. Approval of the primary neonatologist
4. Appropriate caregiver to provide informed consent
5. Is not known to meet or suspected of meeting any of the exclusion criteria (below).

Exclusion Criteria:

1. Participation in another pharmacological intervention trial that involves multiple doses of a medication that may interact with EPO+MLT. Examples of exemptions would include single dose administration for pharmacokinetic studies of an antibiotic, a single or few doses of a new surfactant, or a single intervention to reduce pain.
2. Is on jet ventilator or has not been off jet ventilator for at least 72 hours
3. Has been diagnosed with or is suspected of having a congenital anomaly or genetic disorder associated with brain malformation or life expectancy <40 weeks post menstrual age (PMA). These include but are not limited to TORCH infections associated with radiographic evidence of substantial brain injury, trisomy 13, coarctation of the aorta, and severe liver failure. TORCH infections not associated with radiographic evidence of brain malformation or treatment for presumed TORCH infection are not exclusionary.
4. Is within 3 days of starting treatment for a severe clinical condition which is potentially associated with a life expectancy <3 days. These include but are not limited to disseminated intravascular coagulation (DIC)/severe hematologic crisis, severe sepsis, Hypoxic-ischemic encephalopathy (HIE), severe brain injury
5. Other clinical conditions including:

   Hydrops fetalis Hypertension for age requiring sustained medication Polycythemia (hematocrit >65%)
6. No caregiver to provide consent

The clinical condition of potential candidates will be monitored throughout the eligibility period to ensure the participant's continued candidacy for participating in the trial.

Ages: 12 Hours to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Rate of SAE/DLT including death | 4 weeks after the conclusion of treatment, up to 38 weeks gestational age
  to test the hypothesis that rate of Serious Adverse Events (SAE)/dose limiting toxicity (DLT) with a cocktail of MLT and EPO in very preterm infants with severe intraventricular hemorrhage (sIVH) will have similar rate of SAE/DLT in subjects treated with placebo

SECONDARY OUTCOMES:
Efficacy of EPO plus MLT as assessed by rate of preterm birth related co-morbidities | 4 weeks after the conclusion of treatment, up to 38 weeks gestational age
  Determine whether treatment with EPO plus MLT alters the rate of preterm birth related co-morbidities compared to concurrent placebo controls.

CONTACTS AND LOCATIONS:
Overall Officials: Shenandoah Robinson, MD, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States